CLINICAL TRIAL: NCT01727115
Title: Comparison of Two Extensively Hydrolyzed Formulas for the Treatment of Children With Cow's Milk Intolerance
Brief Title: Althera® Versus Nutramigen / Cow's Milk Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06.04.INF
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NUTRAMIGEN® (Active Comparator): Subjects are orally fed ad libitum (following guidelines printed on the labels).
  Subjects will receive the Nutramigen® formula for a 4 week period
  Then depending of the result of the challenge test we have the following possibilities:
  * If the test is positive: The children continue the formula Nutramigen®
  * If the test is negative: A Follow up formula is given
    * (Nan pro2) if child > 6 months
    * (Nan pro1) if child < 6 months
  Interventions: Other: Infant Formula Feeding
- ALTHERA® (Experimental): Subjects are orally fed ad libitum (following guidelines printed on the labels).
  Subjects will receive the Althera® formula for a 4 week period
  Then depending of the result of the challenge test we have the following possibilities:
  * If the test is positive: The children continue the formula Althera®
  * If the test is negative: A Follow up formula is given
    * (Nan pro2) if child > 6 months
    * (Nan pro1) if child < 6 months
  Interventions: Other: Infant Formula Feeding

INTERVENTIONS:
Other: Infant Formula Feeding — Assigned formula (Althera® or Nutramigen®) for a 4 weeks period.
  * If the challenge is positive: The children continue the assigned formula
  * If the challenge is negative: A Follow up formula is given
    * (Nan pro2) if child > 6 months
    * (Nan pro1) if child < 6 months

SUMMARY:
The primary objective of this study is to demonstrate that ALTHERA® is equal or superior in efficacy than NUTRAMIGEN®

ELIGIBILITY:
Inclusion Criteria:

* Infants from few days of life until 6 months of age
* Birth weight : between 2.500g and 4.500g
* Full term: gestational age between 37 and 42 weeks
* Singleton birth
* Suspicion of a mild/moderate Cow's Milk Proteins Intolerance (CMPI)
* Having obtained the Informed Consent by the Parents or the legal guardian

Exclusion Criteria:

* Exclusive breastfeeding at time of enrolment
* Having been treated before enrolment with an extensively hydrolysed formula
* Disease impairing a normal gut transit (like pyloric stenosis)
* Intolerance to lactose (if already known)
* Receiving an antibiotic treatment at the time of enrolment
* Severe or chronic diarrhea
* Failure to thrive
* Neurologic diseases
* Receiving a medical treatment which could interfere with the protocol or after a surgical intervention
* Infants whose parents / caregivers who cannot be expected to comply with treatment
* Currently participating or having participated in another interventional clinical trial

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome are regurgitations/vomiting, stool consistency, atopic eczema, urticaria and respiratory symptoms after 4 weeks of treatment. | 4 weeks
  regurgitations/vomiting, stool consistency, atopic eczema, urticaria and respiratory symptoms

SECONDARY OUTCOMES:
To assess whether the 2 groups have comparable changes in weight, length and head circumference | 1 year
  weight, length, head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, Professor, Principal Investigator — AZ-Kinderen V.U.B.; Bruno Hauser, Doctor, Principal Investigator — AZ-Kinderen V.U.B.; Thierry Devreker, Doctor, Principal Investigator — AZ-Kinderen V.U.B.; Marc Verghote, Doctor, Principal Investigator — CHR Namur; Christine Halut, Doctor, Principal Investigator — CHR Namur; Olivia Bauraind, Doctor, Principal Investigator — Clinique Saint Pierre; Sandra Mulier, Doctor, Principal Investigator — CHU des Enfants Reine Fabiola; Pascal Lenoir, Doctor, Principal Investigator — Clinique Notre Dame Tournai; Etienne Sokal, Professor, Principal Investigator — Clinique Universitaire Saint Luc; Francoise Smets, Doctor, Principal Investigator — Clinique Universitaire Saint Luc; Francoise Bury, Doctor, Principal Investigator — Clinique de l'Espérance; Stéphanie Colinet, Doctor, Principal Investigator — Clinique de l'Espérance; Stefaan Peeters, Doctor, Principal Investigator — Aalsters Stedelijk ziekenhuis; Patrick Bollen, Doctor, Principal Investigator — AZ Vesalius; Paul Mariën, Doctor, Principal Investigator — Sint Augustinus; Gigi Veereman, Professor, Principal Investigator — Paola Kinderziekenhuis; Myriam VanWinckel, Professor, Principal Investigator — UZ Gent; Jozef Christens, Doctor, Principal Investigator — Maria Ziekenhuis Noord Limburg; Kristien Kamoen, doctor, Principal Investigator — Algemeen Ziekenhuis Maria Middelares; Michèle Scaillon, Doctor, Principal Investigator — CHU des Enfants Reine Fabiola
Locations (14):
- Belgium (14):
  - ASZ, Aalst, Aalst
  - ZNA Middelheim, Antwerp, Antwerp
  - CHU Huderf, Brussels, Brussels Capital
  - AZ VUB, Brussels, Brussels Capital
  - Cliniques Universitaires, Brussels, Brussels Capital
  - Az Maria Middelares, Ghent, Gent
  - UZ Gent Pediatrie, Ghent, Gent
  - Clinique de l'Espérance, Montegnée, Montegnée
  - Centre Hospitalier Regional, Namur, Namur
  - Clinique Saint Pierre, Ottignies, Ottignies
  - Maria Ziekenhuis, Overpelt, Overpelt
  - Az Vesalius, Tongeren, Tongeren
  - CH WAPI Tournai, Tournai, Tournai
  - Sint Augustinus, Wilrijk, Wilrijk

REFERENCES:
- [Derived] Vandenplas Y, Steenhout P, Planoudis Y, Grathwohl D; Althera Study Group. Treating cow's milk protein allergy: a double-blind randomized trial comparing two extensively hydrolysed formulas with probiotics. Acta Paediatr. 2013 Oct;102(10):990-8. doi: 10.1111/apa.12349. Epub 2013 Aug 5. PMID 23837862